CLINICAL TRIAL: NCT03336632
Title: Chidamide Plus Post-transplantation Cyclophosphamide and Cyclosporine to Prevent Graft-versus-host Disease After Myeloablative Conditioning, Matched Peripheral-blood Stem-cell Transplantation
Brief Title: Chidamide Plus PTCy/Cyclosporine to Prevent GVHD After Myeloablative Conditioning, Matched PBSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, MD, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-GVHD-1
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Leukemia, Acute; MDS
Keywords: PBSCT; myeloablative conditioning; HDACi; chidamide
MeSH Terms: conditions — Leukemia | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000; Cyclophosphamide; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide (Experimental): Chidamide, tablets, 5 mg/tablet, 20 mg orally twice weekly from D-7~+14 Cyclophosphamide: 50 mg/Kg intravenously D+3, +4 Cyclosporine A: intravenously then orally 3 mg/Kg D+5~D+100
  Interventions: Drug: Chidamide; Drug: Cyclophosphamide; Drug: cyclosporine A

INTERVENTIONS:
Drug: Chidamide — 20 mg orally, twice weekly from D-7 to D+14
  Other Names: HBI-8000
Drug: Cyclophosphamide — 50 mg/Kg intravenously D+3, +4
Drug: cyclosporine A — 3 mg/Kg intravenously then orally from D+5 to D+100 if no acute graft-versus-host disease
  Other Names: cyclosporine

SUMMARY:
This study is to explore the efficacy and safety of introduction of chidamide in PTCy based GVHD prophylaxis in patients undergoing allogeneic PBSCT.

DETAILED DESCRIPTION:
Eligible patients were aged 16 to 65 years, diagnosed with hematologic malignancy, and had a Karnofsky performance score of ≥70% and were candidates for myeloablative HCT. A 8/8 HLA allelic match between the donor and the recipient at HLA-A, HLA-B, HLA-C, and HLA-DRB1 by high-resolution typing was required. The graft source was PBSC.

Patients received a myeloablative conditioning regimen consisting of oral chidamide given twice weekly at a dose of 20 mg from day -7 to 2 weeks post transplantation, intravenous busulfan 3.2 mg/kg from day -6 to -3, intravenous fludarabine 30 mg/m2 and cytarabine 1g/m2 respectively from day -6 to -2. PBSCs were infused on day 0. GVHD prophylaxis was post-transplantation cyclophosphamide (50 mg/kg on day +3, +4) and cyclosporine (started from day +5). In the absence of GVHD, cyclosporine tapering started on day +100 and discontinued on day +180. Minimal residual disease (MRD) was determined by multi-parameter flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years or older, and ≤ 65 years at time of enrollment
2. Signed informed consent
3. Hematologic disorder requiring allogeneic hematopoietic cell transplantation
4. Left ventricular ejection fraction (LVEF) ≥ 45% by multiple uptake gated acquisition (MUGA) scan or echocardiogram
5. Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and diffusing lung capacity oxygenation (DLCO) adjusted ≥ 50% of predicted values on pulmonary function tests
6. Transaminases (AST, ALT) < 3 times upper limit of normal (ULN) values
7. Creatinine clearance calculated ≥ 50 mL/min
8. Karnofsky Performance Status Score ≥ 60%.
9. Human leukocyte antigen (HLA) matched 8/ (A, B, C, DRB1) related or unrelated donor

Exclusion Criteria:

1. Active infection not controlled with appropriate antimicrobial therapy HIV, hepatitis B (HBcAb positive but HBsAg negative with undetectable viral load are eligible), or hepatitis C infection
2. Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) ≥4
3. Anti-thymocyte globulin (ATG) as part of the conditioning regimen
4. Pregnancy
5. Histone deacetylase (HDAC), DAC, HSP90 inhibitors or valproic acid for the treatment of cancer within 30 days
6. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first chidamide treatment
7. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following: Any history of ventricular fibrillation or torsade de pointes; Bradycardia defined as heart rate (HR)< 45 bpm (Patients with pacemakers are eligible if HR ≥ 45 bpm); Screening electrocardiogram (ECG) with a QTcF > 480 msec; Right bundle branch block + left anterior hemiblock (bifascicular block); Patients with myocardial infarction or unstable angina ≤ 12 months prior to starting study drug; Other clinically significant heart disease (e.g., New York Heart Association (NYHA) class III or IV , uncontrolled hypertension) as per discretion of principal investigator and/or treating physician; Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug with the exception of drugs listed on Appendix B of study documents that are required for hematopoietic cell transplantation (HCT) patients.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
aGVHD | 100 day after infusion of PBSCs
  accumulated incidence of aGVHD

SECONDARY OUTCOMES:
GRFS | 3 years after recruitment
  GVHD free, relapse free survival
DFS | 3 years after recruitment
  Disease free survival
OS | 3 years after recruitment
  Overall survival
cGVHD | 2 yeas after infusion of PBSCs
  accumulated incidence of cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Ting Liu, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No